CLINICAL TRIAL: NCT06113458
Title: Comparing Hypertension Remote Monitoring Evaluation Redesign
Acronym: CHARMED
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P0564385
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard and One-time Training (Active Comparator): Patient level: Standard, automatic reminders Clinic level: One-time training
  Interventions: Behavioral: Standard and One-time Training
- Standard and Practice Facilitation (Experimental): Patient level: Standard, automatic reminders Clinic level: Regular, ongoing coaching
  Interventions: Behavioral: Standard and Practice Facilitation
- High-intensity and One-time Training (Experimental): Patient level: Personalized feedback Clinic level: One-time training
  Interventions: Behavioral: High-intensity and One-time Training
- High-intensity and Practice Facilitation (Experimental): Patient level: Personalized feedback Clinic level: Regular, ongoing coaching
  Interventions: Behavioral: High-intensity and Practice Facilitation

INTERVENTIONS:
Behavioral: Standard and One-time Training — Patient-level intervention: Patients in the standard group will receive automated reminder SMS text messages and remote BP monitoring.
  Clinic-level intervention: Clinics in the one-time training group will receive one-time training on standard work and algorithms, audit and feedback, and panel-based outreach.
  Arms: Standard and One-time Training
Behavioral: Standard and Practice Facilitation — Patient-level intervention: Patients in the standard group will receive automated reminder SMS text messages and remote BP monitoring.
  Clinic-level intervention: Clinics in the practice facilitation group will receive regular/ongoing training on standard work and algorithms, audit and feedback, and panel-based outreach.
  Arms: Standard and Practice Facilitation
Behavioral: High-intensity and One-time Training — Patient-level intervention: Patients in the high-intensity group will receive personalized feedback SMS text messages and remote BP monitoring.
  Clinic-level intervention: Clinics in the one-time training group will receive one-time training on standard work and algorithms, audit and feedback, and panel-based outreach.
  Arms: High-intensity and One-time Training
Behavioral: High-intensity and Practice Facilitation — Patient-level intervention: Patients in the high-intensity group will receive personalized feedback SMS text messages and remote BP monitoring.
  Clinic-level intervention: Clinics in the practice facilitation group will receive regular/ongoing training on standard work and algorithms, audit and feedback, and panel-based outreach.
  Arms: High-intensity and Practice Facilitation

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of evidence-based, adapted, and tailored, patient-focused and clinic-focused strategies to improve blood pressure (BP) control in English- and Spanish-speaking patients with hypertension (HTN).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Any sex/gender
* Any race or ethnicity
* Have hypertension or high blood pressure (BP) (BP >=140/90 mmHg at least twice in the previous 18 months)
* Can read and write English or Spanish
* Be able to provide consent

Exclusion Criteria:

• We will exclude individuals with conditions that might have severe self-management limitations due to a disability or medical condition or might complicate remote BP monitoring, such as self-reported:

* Pregnancy
* Lactating/nursing
* Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in systolic BP (clinic) | Baseline, 6 months
  Clinic-based BP readings in EHR

SECONDARY OUTCOMES:
Change in systolic BP (home) | Baseline, 6 months
  Home-based BP readings
Patient activation and satisfaction | Baseline, 6 months
  Patients will complete the Patient Assessment of Chronic Illness Care (PACIC) survey of 20 questions regarding elements of the care of their chronic condition(s) over the last six months. Patients answer using a Likert scale of answers ranging from 1-5, with 1 signifying "Almost Never" and 5 signifying "Almost Always".
Number of participants with BP control | Baseline, 6 months
  <140/90mmHg, at the patient level within the EHR
Medication intensification when BP is uncontrolled | Baseline, 6 months
  Number of classes of anti-hypertensive medications prescribed per patient
Patient-reported medication adherence | Baseline, 6 months
  Patients will complete the 4-item Krousel-Wood Medication Adherence Scale (M-Wood-MAS-4). The scale score is calculated by summing the points for the 4 questions (scale score ranges from 0 to 4, with higher score indicating worse adherence); low adherence on the K-Wood-MAS-4 is defined as a score ≥1.

CONTACTS AND LOCATIONS:
Overall Officials: Urmimala Sarkar, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyles CR, Khoong EC, Stern RJ, Abtahi N, Sharma AE, Pletcher MJ, Xia F, Garcia F, Shah ND, Tieu L, Sarkar U; CHARMED consortium. Championing Hypertension Remote Monitoring for Equity and Dissemination (CHARMED): A multi-site factorial randomized controlled trial protocol. Contemp Clin Trials. 2025 May;152:107879. doi: 10.1016/j.cct.2025.107879. Epub 2025 Mar 12. PMID 40086748